CLINICAL TRIAL: NCT03835884
Title: First-in-Human Study of the Safety of AR-13503 Sustained Release Intravitreal Implant in Subjects With Neovascular Age-Related Macular Degeneration (nAMD) and Subjects With Diabetic Macular Edema (DME)
Brief Title: A Study Assessing AR-13503 Implant in Subjects With nAMD or DME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AR-13503-CS201
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema
Keywords: Neovascular AMD; Diabetic macular edema; Diabetic retinopathy; Vascular endothelial growth factor; Intravitreal injection
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AR-13503 Implant 10.6 Dose (Experimental): Single dose of AR-13503 Implant 10.6 Dose (10.6 µg) administered as an intravitreal implant into a single eye of up to 6 subjects (3 nAMD and 3 DME) who will be followed for 24 weeks
  Interventions: Drug: AR-13503 Implant 10.6 Dose
- AR-13503 Implant 21.2 Dose (Experimental): Single dose of AR-13503 Implant 21.2 Dose (21.2 µg) administered as intravitreal implants into a single eye of up to 6 subjects (3 nAMD and 3 DME) who will be followed for 24 weeks
  Interventions: Drug: AR-13503 Implant 21.2 Dose
- AR-13503 Implant 42.4 Dose (Experimental): Single dose of AR-13503 Implant 42.4 Dose (42.4 µg) administered as intravitreal implants into a single eye of up to 6 subjects (3 nAMD and 3 DME) who will be followed for 24 weeks
  Interventions: Drug: AR-13503 42.4 Dose
- AR-13503 Implant 63.6 Dose (Experimental): Dose of AR-13503 Implant 63.6 Dose (63.6 µg) administered into a single eye of up to 5 subjects (DME) who will be followed for 24 weeks. Subjects may qualify to receive an additional dose at Week 12.
  Interventions: Drug: AR-13503 63.6 Dose

INTERVENTIONS:
Drug: AR-13503 Implant 10.6 Dose — AR-13503 Implant 10.6 Dose (10.6 µg) administered as an intravitreal implant into a single eye
  Arms: AR-13503 Implant 10.6 Dose
Drug: AR-13503 Implant 21.2 Dose — AR-13503 Implant 21.2 Dose (21.2 µg) administered as intravitreal implants into a single eye
  Arms: AR-13503 Implant 21.2 Dose
Drug: AR-13503 42.4 Dose — AR-13503 Implant 42.4 Dose (42.4 µg) administered as intravitreal implants into a single eye
  Arms: AR-13503 Implant 42.4 Dose
Drug: AR-13503 63.6 Dose — AR-13503 Implant 63.6 Dose (63.6 µg) administered as intravitreal implants into a single eye
  Arms: AR-13503 Implant 63.6 Dose

SUMMARY:
First-in-Human Study of the Safety of AR-13503 Sustained Release Intravitreal Implant in Subjects with Neovascular Age-Related Macular Degeneration (nAMD) and Subjects with Diabetic Macular Edema (DME)

DETAILED DESCRIPTION:
This is a first-in-human study conducted in 2 sequential stages; each stage is 24 weeks in duration. Subjects with nAMD and subjects with DME were evaluated in Stage 1. Subjects with DME will be evaluated in Stage 2.

ELIGIBILITY:
Inclusion Criteria for Subjects with Neovascular Age-Related Macular Degeneration (nAMD)

1. 50 years of age or older
2. Presence of active subfoveal or juxtafoveal Choroidal Neovascularization (CNV) (any subtype) with leakage affecting the fovea secondary to Age-Related Macular Degeneration (AMD)
3. Best Corrected Visual Acuity (BCVA) in the study eye at Baseline (Day 0):

   Stage 1: between 65 and 10 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (20/50 and 20/640 Snellen equivalent)
4. Able and willing to give signed informed consent and follow study instructions

Inclusion Criteria for Subjects with Diabetic Macular Edema (DME)

Subjects with Diabetic Macular Edema (DME) must meet all the following criteria to enter into the study:

1. 18 years of age or older
2. Type 1 or 2 diabetes mellitus with center-involved DME
3. BCVA in the study eye at Baseline (Day 0):

   Stage 1: between 65 and 10 ETDRS letters (20/50 and 20/640 Snellen equivalent) Stage 2: between 70 and 20 ETDRS letters (20/40 and 20/400 Snellen equivalent)
4. Able and willing to give signed informed consent and follow study instructions

Exclusion Criteria for Subjects with Neovascular Age-Related Macular Degeneration (nAMD)

Ophthalmic:

1. Use of intravitreal aflibercept within 8 weeks, ranibizumab or bevacizumab within 6 weeks
2. History of vitreoretinal surgery in the study eye
3. Any ocular disease in the study eye that in the Investigator and Reading Center's opinion may confound assessment of the macula, affect central vision, confound results, or preclude improvement in visual acuity
4. Any current or history of periocular or intraocular inflammation or evidence of infection in either eye
5. Media clarity insufficient to obtain quality fundus and OCT images in the study eye

Systemic:

1. History or current systemic condition that in the Investigator opinion preclude the safe administration of the study treatment or confound results
2. History of allergy or sensitivity to fluorescein or povidone iodine
3. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control
4. Participation in an investigational study within 30 days of Screening

Exclusion Criteria for Subjects with DME

Ophthalmic:

1. Use of intraocular or periocular corticosteroids within 6 months, aflibercept within 8 weeks, ranibizumab or bevacizumab within 6 weeks
2. History of vitreoretinal surgery in the study eye
3. High risk proliferative diabetic retinopathy in the study eye and related complications
4. Structural damage to the center or the macula that is likely to preclude improvement in visual acuity in the study eye after resolution of the DME
5. Media clarity insufficient to obtain quality fundus and OCT images in the study eye

Systemic:

1. History or current medical condition that in the Investigator's opinion preclude the safe administration of the study treatment or confound results
2. History of allergy or sensitivity to fluorescein or povidone iodine
3. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control
4. Participation in an investigational study within 30 days of Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Number of ocular and non-ocular TEAEs | 24 weeks
  Number of ocular and non-ocular treatment-emergent adverse events (TEAEs), summarized at the subject level by system organ class and preferred term, and also by severity and relatedness to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kerr, Study Director — Aerie Pharmaceuticals, Inc.
Locations (6):
- United States (6):
  - Retinal Research Institute, LLC, Gilbert, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Sterling Vision, PC dba Oregon Retina, Eugene, Oregon
  - Valley Retina Institute, P.A., Harlingen, Texas
  - Medical Center Ophthamology Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No